CLINICAL TRIAL: NCT03841526
Title: Phase 2 Randomized Placebo-Controlled Double-Blind Parallel Study to Evaluate Glucagon RTU (Glucagon Injection) Compared to Standard of Care for Prevention of Exercise-Induced Hypoglycemia During Regular Aerobic Exercise in Adults With T1D
Brief Title: Glucagon Ready-to-Use (RTU) for Prevention of Exercise-Induced Hypoglycemia During Aerobic Exercise in Adults With T1D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XSMP-204
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hypoglycemia
Keywords: Exercise; Glucagon; Insulin
MeSH Terms: conditions — Hypoglycemia; Motor Activity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: CRC Phase: randomized, placebo-controlled, double-blind, two-treatment, two-period, crossover comparison in a clinical research center (CRC) setting. The subjects were re-randomized into the Outpatient Phase: randomized, placebo-controlled, partially double-blind, 3-arm parallel comparison in an outpatient setting.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: CRC Phase was a fully masked double-blind crossover with each subject receiving each treatment 1 time. In the Outpatient Phase, the two arms with 50% insulin pump reduction were double-blind (fully masked) and the arm with Glucagon RTU and no insulin pump reduction was open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CRC Phase: Glucagon RTU With Insulin Pump Reduction (Experimental): CRC Phase: 2-arm randomized double-blind crossover, Glucagon RTU Injection 30 microliters of 0.15 mg injection with 50% reduction in the insulin pump
  Interventions: Drug: Glucagon RTU Injection With Insulin Pump Reduction
- CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction (Placebo Comparator): CRC Phase: 2-arm randomized double-blind crossover, Vehicle for Glucagon RTU Injection 30 microliters vehicle with 50% reduction in the insulin pump
  Interventions: Other: Vehicle for Glucagon RTU Injection With Insulin Pump Reduction
- Outpatient Phase: Glucagon RTU With Insulin Pump Reduction (Experimental): Outpatient Phase: 3-arm randomized comparison (2-arm double-blind, 1-arm open-label), Glucagon RTU Injection 30 microliters of 0.15 mg injection with 50% reduction in the insulin pump (double-blind arm)
  Interventions: Drug: Glucagon RTU Injection With Insulin Pump Reduction
- Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction (Placebo Comparator): Outpatient Phase: 3-arm randomized comparison (2-arm double-blind, 1-arm open-label), Vehicle for Glucagon RTU Injection 30 microliters vehicle with 50% reduction in the insulin pump (double-blind arm)
  Interventions: Other: Vehicle for Glucagon RTU Injection With Insulin Pump Reduction
- Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction (Experimental): Outpatient Phase: 3-arm randomized comparison (2-arm double-blind, 1-arm open-label), Glucagon RTU Injection 30 microliters of 0.15 mg injection without a reduction in the insulin pump (open-label arm)
  Interventions: Drug: Glugaon RTU Injection Without Insulin Pump Reduction

INTERVENTIONS:
Drug: Glucagon RTU Injection With Insulin Pump Reduction — 0.15 mg injection with 50% pump reduction
  Other Names: XP-3994
  Arms: CRC Phase: Glucagon RTU With Insulin Pump Reduction; Outpatient Phase: Glucagon RTU With Insulin Pump Reduction
Other: Vehicle for Glucagon RTU Injection With Insulin Pump Reduction — vehicle injection with 50% pump reduction
  Other Names: Placebo
  Arms: CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction; Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction
Drug: Glugaon RTU Injection Without Insulin Pump Reduction — 0.15 mg injection without pump reduction
  Other Names: XP-3994
  Arms: Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, 2-treatment, 2-period, crossover comparison in a clinical research center (CRC) setting, followed by a randomized, placebo-controlled, double-blinded, 2-arm parallel comparison with a third open-label arm in an outpatient setting. The purpose of the study is to evaluate the preliminary efficacy and safety of Glucagon Ready-to-Use [RTU] to prevent exercise-induced hypoglycemia (EIH) in adults with Type 1 diabetes mellitus (T1D), who perform regular, moderate-to-high intensity aerobic exercise.

DETAILED DESCRIPTION:
There were 2 phases of this study: CRC and Outpatient. The initial posting of this study reflected the 3 treatment arms included in the Outpatient Phase of the study, without including the CRC and Outpatient Phases separately.

CRC Phase:

The CRC Phase was comprised of 2 visits that included daytime exercise sessions at the CRC or a comparable setting. Subjects were randomized to receive their first treatment at Visit 3 and crossed over (2 to 28 day washout) to their second treatment at Visit 4. The treatments were a single treatment with 30 microliters of either Glucagon RTU (0.15 mg) or placebo with a 50% insulin pump reduction. Blood glucose was assessed 15 minutes prior to the start of exercise, at the start of exercise, and then 15, 30, 45, 60, and 75 minutes from the start of exercise.

Outpatient Phase:

After completion of the CRC Phase, subjects entered the 12-week Outpatient Phase. Subjects were to maintain a weekly exercise average of 2 to 3 sessions of at least 30 minutes duration. Subjects were assigned randomly in 1:1:1 ratio to administer 30 microliters of one of the following prior to the exercise sessions: Glucagon RTU (0.15 mg) with a 50% insulin pump reduction, placebo with a 50% pump reduction or Glucagon RTU (0.15 mg) without an insulin pump reduction. Blood glucose was assessed 15 minutes prior to the start of exercise, just before exercise, after 30 minutes of exercise, at the end of exercise (if longer than 30 minutes), and 30 minutes post-exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of presumed autoimmune type 1 diabetes, receiving daily insulin via continuous subcutaneous insulin infusion.
2. Age 18 to < 65 years.
3. Duration of type 1 diabetes ≥ 2 years.
4. Random C-peptide < 0.6 ng/mL (<198 pmol/L).
5. Using insulin therapy by continuous subcutaneous insulin infusion pump for at least 6 months.
6. History of exercise-related hypoglycemia.
7. Performs aerobic exercise regularly (2-3 times per week), and desires to exercise per American Diabetes Association guidelines (150 minutes per week). Examples of aerobic exercise include: power walking, hiking, running/jogging, cycling, swimming, cross country skiing, and aerobic fitness classes.
8. Will abstain from the use of non-insulin diabetes therapies such as sodium glucose co-transporter 2, glucagon like peptide-1, and metformin for the duration of the study.
9. Subject must be willing to adhere to the protocol requirements for the duration of the study.
10. Subject has provided informed consent as evidenced by a signed/dated informed consent form completed before any trial-related activities occur.

Exclusion Criteria:

1. Frequently experience hyperglycemia with exercise, in the clinical judgement of the investigator.
2. Pregnant and/ or Nursing: For female subjects of childbearing potential, there is a requirement for a negative urine pregnancy test and for agreement to use contraception and to refrain from breast feeding during the study, and for at least 1 week after the last dose of study drug. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intra-uterine device, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
3. One or more severe hypoglycemic episodes in the past 12 months (as defined by an episode that required third party assistance for treatment).
4. Uses inhaled insulin.
5. Hemoglobin A1c > 9.0% at Screening.
6. Renal insufficiency (serum creatinine greater than 3 mg/dL (0.17 mmol/L)).
7. Serum alanine aminotransferase or aspartate aminotransferase equal to or greater than 3 times the upper limit of normal.
8. Hepatic synthetic insufficiency as defined as a serum albumin of less than 3 mg/dL (0.17 mmol/L); or serum bilirubin greater than 2 mg/dL (0.11 mmol/L).
9. Hematocrit of less than or equal to 30%.
10. Mean of triplicate blood pressure (BP) readings at Screening where systolic BP <90 or >150 mm Hg, or diastolic BP <50 or >100 mm Hg.
11. Clinically significant electrocardiogram abnormalities.
12. Use of > 2.0 U/kg total insulin dose per day.
13. Inadequate bilateral venous access in both arms.
14. Congestive heart failure, New York Heart Association class III or IV.
15. Active malignancy within 5 years from Screening, except basal cell or squamous cell skin cancers.
16. Major surgical operation within 90 days prior to screening, or planned surgical operation during the study.
17. History of seizure disorders.
18. Bleeding disorder, treatment with warfarin or any anticoagulants, or platelet count below 50,000 mm3 at Screening.
19. History of pheochromocytoma or disorder with increased risk of pheochromocytoma (multiple endocrine neoplasia type 2, neurofibromatosis, or Von Hippel-Lindau disease).
20. History of insulinoma.
21. History of allergies to glucagon or glucagon-like products, or any history of significant hypersensitivity to glucagon or any related products or to any of the excipients (dimethylsulfoxide, mannitol, & trehalose) in the investigational formulation.
22. History of glycogen storage disease.
23. Subject tests positive for human immunodeficiency virus, hepatitis C virus, or active hepatitis B virus infection at Screening.
24. Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
25. Active substance or alcohol abuse, in the opinion of the investigator. Subjects reporting active marijuana use or testing positive for tetrahydrocannabinol via rapid urine test will be allowed to participate in the study at the discretion of the investigator.
26. Participation in other studies involving administration of an investigational therapeutic agent (drug or device) within 30 days or 5 half-lives, whichever is longer, before Screening for the current study and during participation in the current study.
27. Any reason the investigator deems exclusionary.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Junaidi, MD, Study Chair — Xeris Pharmaceuticals
Locations (1):
- LMC Clinical Research Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aronson R, Riddell MC, Conoscenti V, Junaidi MK. Effect of Mini-Dose Ready-to-Use Liquid Glucagon on Preventing Exercise-Associated Hypoglycemia in Adults With Type 1 Diabetes. Diabetes Care. 2023 Apr 1;46(4):765-772. doi: 10.2337/dc22-1145. PMID 36689626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 48 subjects to participate in the study with a CRC phase followed by an Outpatient phase. The 45 subjects that completed the CRC phase were re-randomized prior to entering the Outpatient phase of the study.
Groups:
- CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction: CRC Phase (2-arm randomized double-blind crossover): Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump to Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump to Outpatient Phase (3-arm randomized comparison, 2-arm double-blind, 1-arm open-label): Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump (double-blind arm)
- CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Vehicle With 50% Reduction: CRC Phase (2-arm randomized double-blind crossover): Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump to Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump to Outpatient Phase (3-arm randomized comparison, 2-arm double-blind, 1-arm open-label): Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump (double-blind arm)
- CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU Without Reduction: CRC Phase (2-arm randomized double-blind crossover): Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump to Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump to Outpatient Phase (3-arm randomized comparison, 2-arm double-blind, 1-arm open-label): Glucagon RTU Injection 0.15 mg injection without reduction in the insulin pump (open-label arm)
- CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction: CRC Phase (2-arm randomized double-blind crossover): Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump to Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump to Outpatient Phase (3-arm randomized comparison, 2-arm double-blind, 1-arm open-label): Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump (double-blind arm)
- CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Vehicle With 50% Reduction: CRC Phase (2-arm randomized double-blind crossover): Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump to Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump to Outpatient Phase (3-arm randomized comparison, 2-arm double-blind, 1-arm open-label): Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump (double-blind arm)
- CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU Without Reduction: CRC Phase (2-arm randomized double-blind crossover): Vehicle for Glucagon RTU Injection with 50% reduction in the insulin pump to Glucagon RTU Injection 0.15 mg injection with 50% reduction in the insulin pump to Outpatient Phase (3-arm randomized comparison, 2-arm double-blind, 1-arm open-label): Glucagon RTU Injection 0.15 mg injection without reduction in the insulin pump (open-label arm)
Period: CRC Phase: First Treatment
Arm/Group | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Vehicle With 50% Reduction | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU Without Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Vehicle With 50% Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU Without Reduction
Started | 8 | 10 | 6 | 11 | 5 | 8
Received 1st CRC Dose | 8 | 10 | 6 | 11 | 5 | 8
Completed | 8 | 10 | 6 | 11 | 5 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: CRC Phase: Second Treatment
Arm/Group | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Vehicle With 50% Reduction | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU Without Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Vehicle With 50% Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU Without Reduction
Started | 8 | 10 | 6 | 11 | 5 | 8
Received 2nd CRC Dose | 7 | 10 | 6 | 9 | 5 | 8
Completed | 7 | 10 | 6 | 9 | 5 | 8
Not Completed | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Outpatient Phase Treatment
Arm/Group | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Vehicle With 50% Reduction | CRC: Glucagon RTU to Vehicle With 50% Reduction to Outpatient: Glucagon RTU Without Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU With 50% Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Vehicle With 50% Reduction | CRC: Vehicle to Glucagon RTU With 50% Reduction to Outpatient: Glucagon RTU Without Reduction
Started | 7 | 10 | 6 | 9 | 5 | 8
Received at Least 1 Outpatient Dose | 7 | 9 | 6 | 9 | 5 | 8
Completed | 7 | 9 | 5 | 9 | 5 | 7
Not Completed | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline information is presented for the Safety population for the CRC Phase (Period 1) of the study, this includes all randomized subjects who received at least one dose of study drug.
Groups:
- Glucagon RTU Crossover to Placebo: CRC Stage: Glucagon RTU to Placebo Crossover Group (Glucagon RTU Injection 30 microliters of 0.15 mg injection crossover to vehicle injection of 30 microliters) with 50% reduction in the insulin pump
- Placebo Crossover to Glucagon RTU: CRC Stage: Placebo to Glucagon RTU Crossover Group (vehicle injection of 30 microliters crossover to Glucagon RTU Injection 30 microliters of 0.15 mg injection) with 50% reduction in the insulin pump
- Total: Total of all reporting groups
Arm/Group | Glucagon RTU Crossover to Placebo | Placebo Crossover to Glucagon RTU | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.47) | 34.7 (10.54) | 37.3 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 24 | 22 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 20 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
Weight [Mean (Standard Deviation); unit: kg] | 82.15 (16.344) | 75.91 (16.769) | 79.03 (16.681)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.051 (4.6277) | 26.515 (4.7469) | 26.783 (4.6454)

OUTCOME MEASURES:

1. Primary Outcome: Outpatient Phase: Incidence Rate of Hypoglycemia During and After Moderate to High Intensity Aerobic Exercise.
Description: Mean incidence rate of hypoglycemia during and after sessions of moderate to high intensity aerobic exercise in 12-week Outpatient Phase. Incidence rate is defined as the number of hypoglycemic events divided by the total number of qualified exercise sessions, assessed at group level.
  Qualified exercise session is: (1) confirmed blood glucose of 100-180 mg/dL prior to start of exercise, (2) self-administered study drug no more than 10 min prior to exercise (5 min target), (3) conducted a protocol allowed exercise of moderate to high intensity for at least 30 min and no longer than 75 min, and (4) achieved a target heart rate of 80% of maximum calculated heart rate at least once during session.
  Exercise sessions were to occur at least 2-3 times per week. Only 1 qualified exercise session/subject/day was included in the analysis (the first if >1).
  Hypoglycemic event defined as any hypoglycemic event occurring within 30 (+2) min after completion of a qualified exercise session.
Time Frame: Daily; During the 12-week Outpatient Phase qualified exercise sessions were assessed daily and associated hypoglycemia events were assessed continuously during and within the 30 (+2) minute period following a qualified exercise session.
Population: All randomized subjects in the Outpatient Phase with data.
Measure: Number; unit: events/session
Groups:
- Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction: Outpatient Phase: 3-arm randomized comparison (2-arm double-blind, 1-amr open-label), Glucagon RTU Injection 30 microliters of 0.15 mg injection without a reduction in the insulin pump (open-label arm)
- Outpatient Phase: Overall: All 3 treatment groups in the Outpatient Phase
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction | Outpatient Phase: Overall
Number analyzed (Participants) | 16 | 14 | 14 | 44
events/session | 0.12 | 0.39 | 0.16 | 0.24
Statistical Analysis 1: Comparison: Outpatient Phase: Glucagon RTU With Insulin Pump Reduction vs Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction vs Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction; The primary efficacy analysis was analyzed by analysis of variance (ANOVA) comparing the mean incidence rates among the 3 treatment groups in the Outpatient Phase. If the performed Friedman's test yielded an overall p-value less than 0.05, post-hoc analysis of groups means were conducted to statistically determine which group means differed; Test type: Other — Parameters that did not meet normality criterion were analyzed non-parametrically. Overall treatment effect was assessed using Friedman's test; p = 0.0002, ANOVA
Statistical Analysis 2: Comparison: Outpatient Phase: Glucagon RTU With Insulin Pump Reduction vs Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction; If the overall treatment effect was significant, pairwise treatment comparisons were assessed using: If a difference between 2 treatments was normally distributed, the Tukey Test was used or if not normally distributed and the distribution was highly skewed, the sign test/Kruskal-Allis test was used; Test type: Other; p < 0.0001, Tukey Test/Kruskal-Wallis Test; Tukey Test (if the difference between 2 treatments was normally distributed) or Kruskal-Wallis Test (if not normally distributed)
Statistical Analysis 3: Comparison: Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction vs Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.0032, Tukey Test/Kruskal-Wallis Test; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Outpatient Phase: Glucagon RTU With Insulin Pump Reduction vs Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.2072, Tukey Test/Kruskal-Wallis Test; [statistical method as in outcome 1, analysis 2]

2. Primary Outcome: Outpatient Phase: Mean Number of Hypoglycemic Events
Description: Outpatient Phase: Mean number of hypoglycemic events associated with the qualified exercise sessions, assessed at group level.
  A qualified exercise session was defined as one were (1) a confirmed blood glucose value of 100-180 mg/dL prior to start of exercise, (2) self-administered the study drug no more than 10 minutes prior to exercise (5 minutes was the target), (3) conducted a protocol allowed exercise for moderate to high intensity for at least 30 minutes and no longer than 75 minutes, and (4) achieved a target heart rate of 80% of maximum calculated heart rate at least once during the session.
  A hypoglycemic event was defined as any hypoglycemic event occurring during or within 30 (+2) minutes after completion of a qualified exercise session.
  Exercise sessions were expected to occur at least 2 to 3 times per week. Only 1 qualified exercise session per subject per day was included in the analysis (the first if >1).
Time Frame: Daily; During the 12-week Outpatient Phase qualified exercise sessions were assessed daily and associated hypoglycemia events were assessed continuously throughout the 30 (+2) minute period following a qualified exercise session.
Population: All randomized subjects in the Outpatient Phase with data.
Measure: Number; unit: mean number of events/participant
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction | Outpatient Phase: Overall
Number analyzed (Participants) | 16 | 14 | 14 | 44
mean number of events/participant | 1.94 | 8.43 | 2.86 | 4.3

3. Primary Outcome: Outpatient Phase: Mean Number of Qualified High Intensity Aerobic Exercise Sessions
Description: Outpatient Phase: Mean number of qualified exercise sessions, assessed at group level.
  A qualified exercise session was defined as one were (1) a confirmed blood glucose value of 100-180 mg/dL prior to start of exercise, (2) self-administered the study drug no more than 10 minutes prior to exercise (5 minutes was the target), (3) conducted a protocol allowed exercise for moderate to high intensity for at least 30 minutes and no longer than 75 minutes, and (4) achieved a target heart rate of 80% of maximum calculated heart rate at least once during the session.
  Exercise sessions were expected to occur at least 2 to 3 times per week. Only 1 qualified exercise session per subject per day was included in the analysis (the first if >1).
Time Frame: Daily; During the 12-week Outpatient Phase the occurrence of qualified exercise sessions were assessed daily.
Population: All randomized subjects in the Outpatient Phase with data.
Measure: Number; unit: mean number of sessions/participant
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction | Outpatient Phase: Overall
Number analyzed (Participants) | 16 | 14 | 14 | 44
mean number of sessions/participant | 15.69 | 21.64 | 17.36 | 18.11

4. Secondary Outcome: CRC Phase: Interstitial Glucose Below Target Range
Description: Analysis of interstitial glucose (IG) was performed by treatment, independent of the order of treatment during the randomized cross-over CRC Phase. The number of participants are categorized by the following IG levels:
  Below range, as defined by IG <= 70 mg/dl (<=3.89 mmol/L); Between range, as defined by IG between 54 to 70 mg/dL (3 to 3.89 mmol/L); Below range, as defined by IG <54 mg/dL (<3 mmol/L)
Time Frame: Visit 3 (Day 1) and Visit 4 (Day 3 or any day up to Day 29); Assessed continuously 0-300 minutes following the start of the exercise session corresponding to each of the treatments during the corresponding in-clinic visit during the CRC Phase.
Population: All randomized subjects in the CRC phase.
Measure: Count of Participants; unit: Participants
Groups:
- CRC Phase: Glucagon RTU With Insulin Pump Reduction: CRC Phase: 2-arm randomized double-blind crossover, Glucagon Ready To Use (RTU) Injection 30 microliters of 0.15 mg injection with 50% reduction in the insulin pump.
  Glucagon RTU Injection With Insulin Pump Reduction: 0.15 mg injection with 50% pump reduction
- CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction: CRC Phase: 2-arm randomized double-blind crossover, Vehicle for Glucagon Ready To Use (RTU) Injection 30 microliters vehicle with 50% reduction in the insulin pump.
  Vehicle for Glucagon RTU Injection With Insulin Pump Reduction: vehicle injection with 50% pump reduction
- CRC Phase: Overall: CRC Phase: Glucagon RTU and/or Vehicle 30 microliters with 50% reduction in insulin pump
Arm/Group | CRC Phase: Glucagon RTU With Insulin Pump Reduction | CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | CRC Phase: Overall
Number analyzed (Participants) | 48 | 48 | 48
Participants
  Below range (<=70 mg/dL) | 4 | 5 | 9
  Between range (54-70 mg/dL) | 4 | 5 | 9
  Below range (<54 mg/dL) | 1 | 1 | 2
Statistical Analysis 1: Comparison: CRC Phase: Glucagon RTU With Insulin Pump Reduction vs CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction; Test type: Other; p = 1.0000, Fisher Exact

5. Secondary Outcome: Outpatient Phase: Interstitial Glucose Levels Below Target Range
Description: Analysis of interstitial glucose (IG) was performed by treatment, during the randomized Outpatient Phase. The number of participants are categorized by the following IG levels:
  Below range, as defined by IG <= 70 mg/dl (<=3.89 mmol/L); Between range, as defined by IG between 54 to 70 mg/dL (3 to 3.89 mmol/L); Below range, as defined by IG <54 mg/dL (<3 mmol/L)
Time Frame: Visit 3 (Day 1) and Visit 4 (Day 3 or any day up to Day 29); Assessed continuously 0-300 minutes following the start of each qualified exercise session corresponding to each of the treatments during the Outpatient Phase.
Population: All randomized subjects in the Outpatient Phase with data.
Measure: Count of Participants; unit: Participants
Groups:
- Outpatient Phase: Overall: Outpatient Phase: All subjects across the 3 treatment arms in the Outpatient Phase.
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction | Outpatient Phase: Overall
Number analyzed (Participants) | 16 | 15 | 14 | 45
Participants
  Below range <=70 mg/dL | 14 | 14 | 12 | 40
  Between Range 54-70 mg/dL | 14 | 14 | 12 | 40
  Below range <54 mg/dL | 11 | 14 | 9 | 34
Statistical Analysis 1: Comparison: Outpatient Phase: Glucagon RTU With Insulin Pump Reduction vs Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction; Test type: Other; p = 0.8590, Chi-squared

6. Secondary Outcome: Outpatient Phase: Insulin Use Change From Baseline
Description: Insulin use as reported by subject as Change from Outpatient Phase Baseline at Study Weeks 4, 8, and 12
Time Frame: Insulin use measured continuously from Study Baseline to End of Study and assessed during Outpatient Phase as Change from Outpatient Phase Baseline at Study Weeks 4, 8, and 12
Population: All randomized subjects in the Outpatient Phase with change from Outpatient Phase Baseline data available at Study Weeks 4, 8, and 12
Measure: Mean (Standard Deviation); unit: units of insulin
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction
Number analyzed (Participants) | 11 | 12 | 7
units of insulin
  Fiasp (Insluin Aspart) - Change from Baseline at Week 4: number analyzed (Participants) | 1 | 2 | 1
  Fiasp (Insluin Aspart) - Change from Baseline at Week 4 | -2.80 | 2.60 (0.141) | 0.10
  Fiasp (Insluin Aspart) - Change from Baseline at Week 8: number analyzed (Participants) | 0 | 3 | 0
  Fiasp (Insluin Aspart) - Change from Baseline at Week 8 |  | -2.10 (1.353) |
  Fiasp (Insluin Aspart) - Change from Baseline at Week 12: number analyzed (Participants) | 1 | 2 | 0
  Fiasp (Insluin Aspart) - Change from Baseline at Week 12 | -7.60 | -1.70 (4.808) |
  Humalog (Insulin Lispro) - Change from Baseline at Week 4: number analyzed (Participants) | 0 | 2 | 1
  Humalog (Insulin Lispro) - Change from Baseline at Week 4 |  | 3.05 (1.909) | 6.20
  Humalog (Insulin Lispro) - Change from Baseline at Week 8: number analyzed (Participants) | 1 | 1 | 2
  Humalog (Insulin Lispro) - Change from Baseline at Week 8 | 0.90 | 7.20 | 3.20 (9.758)
  Humalog (Insulin Lispro) - Change from Baseline at Week 12: number analyzed (Participants) | 1 | 2 | 4
  Humalog (Insulin Lispro) - Change from Baseline at Week 12 | 0.60 | 1.05 (3.041) | -0.85 (5.498)
  NovoRapid (Insulin Aspart) - Change from Baseline at Week 4: number analyzed (Participants) | 4 | 3 | 2
  NovoRapid (Insulin Aspart) - Change from Baseline at Week 4 | -2.43 (1.559) | -1.57 (2.558) | -2.85 (3.041)
  NovoRapid (Insulin Aspart) - Change from Baseline at Week 8: number analyzed (Participants) | 4 | 4 | 0
  NovoRapid (Insulin Aspart) - Change from Baseline at Week 8 | -0.15 (3.901) | -2.85 (3.834) |
  NovoRapid (Insulin Aspart) - Change from Baseline at Week 12: number analyzed (Participants) | 4 | 1 | 0
  NovoRapid (Insulin Aspart) - Change from Baseline at Week 12 | -0.05 (10.872) | -4.20 |

7. Secondary Outcome: Outpatient Phase: Barriers to Physical Activity Diabetes (Type 1): BAPAD-1 Change From Baseline
Description: Change from Baseline to End of the Outpatient Phase in Score on Barriers to Physical Activity in Type 1 Diabetes (BAPAD-1) Questionnaire A total of 12 factors were scored from 1=unlikely (min.) to 7=extremely likely (max.) for their propensity to keep the subject from practicing regular physical exercise during the next 6 months. Lower scores are considered better, while higher scores are considered worse outcomes. The higher the score (1 to 7), the less likely the subject was to engage in exercise.
  The mean of the scores of the 12 factors were calculated for each subject and the overall mean for the subjects was calculated at a group level with overall mean and standard deviation calculated at Baseline (Visit 3) and Follow-up/Early Termination (Visit 11) to calculate change from Baseline. Subject level and overall means could range from 1 to 7.
Time Frame: Baseline to End of Study measured at Outpatient Phase Baseline (Visit 3, Day 1) and Follow-up (Visit 11, 14-21 days after last exercise session, up to Day 134) or Early Termination (at time of discontinuation)
Population: All randomized subjects in the Outpatient Phase with data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction
Number analyzed (Participants) | 16 | 15 | 14
score on a scale
  Baseline BAPAD-1 (Study Visit 3) | 2.25 (0.894) | 2.17 (0.857) | 2.59 (0.957)
  Change from Baseline at Follow-up in BAPAD-1 (Study Visit 11): number analyzed (Participants) | 15 | 13 | 12
  Change from Baseline at Follow-up in BAPAD-1 (Study Visit 11) | 0.01 (0.988) | -0.38 (0.781) | -0.34 (0.890)
  Change from Baseline at Early Termination in BAPAD-1: number analyzed (Participants) | 0 | 0 | 2
  Change from Baseline at Early Termination in BAPAD-1 |  |  | -1.00 (0.141)

8. Secondary Outcome: Outpatient Phase: HFS-II Overall Score Change From Baseline
Description: Change from Baseline in Score on Hypoglycemia Fear Survey-II (HFS-II)
  A total of 33 items were scored from 0=never (min.) to 4=almost always (max.) for how often in the past 6 months they had done the following:
  Behavior (15 items): things that people with diabetes often do to avoid low blood sugar.
  Worry (18 items): things that people with diabetes often worry about because of low blood sugar.
  Lower scores are considered better outcomes, higher scores are considered worse outcomes.
  The higher the score (0 to 4), the greater the subject's fear of hypoglycemia. The mean of the scores of the 33 items were calculated for each subject and the overall mean for the subjects was calculated at a group level with overall mean and standard deviation calculated at Baseline (Visit 3) and Follow-up/Early Termination (Visit 11) to calculate change from Baseline. Subject level and overall means could range from 0 to 4.
Time Frame: as for outcome 7
Population: All randomized subjects in the Outpatient Phase with data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction
Number analyzed (Participants) | 16 | 15 | 14
score on a scale
  Baseline | 1.28 (0.293) | 1.16 (0.479) | 1.50 (0.746)
  Change from Baseline at Follow-up (Visit 11): number analyzed (Participants) | 15 | 13 | 12
  Change from Baseline at Follow-up (Visit 11) | -0.19 (0.424) | -0.01 (0.290) | -0.03 (0.280)
  Change from Baseline at Early Termination: number analyzed (Participants) | 0 | 0 | 2
  Change from Baseline at Early Termination |  |  | -0.60 (0.849)

9. Secondary Outcome: Outpatient Phase: Hypoglycemic Confidence Scale (HCS) Change From Baseline
Description: Change from Baseline in Score on Hypoglycemia Confidence Scale (HCS)
  The 9-item scale assessed a subject's confidence about safety regarding hypoglycemia. The questionnaire had 4 responses possible for each question, ranging from 1=not confident at all (min.) to 4=very confident (max.). Higher scores are considered better outcomes, while lower scores are considered worse outcomes. The lower the score (1 to 4), the less likely the subject was to engage in exercise.
  The mean of the scores of the 9 items were calculated for each subject and the overall mean for the subjects was calculated at a group level with overall mean and standard deviation calculated at Baseline (Visit 3) and Follow-up/Early Termination (Visit 11) to calculate change from Baseline. Subject level and overall means could range from 1 to 4.
Time Frame: as for outcome 7
Population: All randomized subjects in the Outpatient Phase with data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Glucagon RTU Without Insulin Pump Reduction: Outpatient Phase: 3-arm randomized comparison (2-arm double-blind, 1-arm open-label), Glucagon RTU Injection 30 microliters of 0.15 mg injection without a reduction in the insulin pump (open-label arm)
Arm/Group | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Glucagon RTU Without Insulin Pump Reduction
Number analyzed (Participants) | 16 | 15 | 14
score on a scale
  Baseline | 3.23 (0.541) | 3.34 (0.616) | 3.20 (0.447)
  Change from Baseline at Follow-up (Visit 11): number analyzed (Participants) | 15 | 13 | 12
  Change from Baseline at Follow-up (Visit 11) | 0.07 (0.413) | 0.17 (0.298) | 0.20 (0.357)
  Change from Baseline at Early Termination: number analyzed (Participants) | 0 | 0 | 2
  Change from Baseline at Early Termination |  |  | 0.15 (0.778)

10. Other Pre Specified Outcome: CRC Phase: Incidence Rate of Hypoglycemia During and After Moderate to High Intensity Aerobic Exercise Exercise.
Description: Mean incidence rate of hypoglycemia during or after moderate to high intensity aerobic exercise at each CRC Phase visit. With crossover, each subject had 2 exercise sessions; 1 visit and exercise session with each treatment (the combined data are presented in the Overall category) and assessed at the group level.
  Incidence rate is defined as the number of hypoglycemic events divided by the total number of qualified exercise sessions, assessed at group level.
  Qualified exercise session is: (1) confirmed blood glucose of 100-180 mg/dL prior to start of exercise, (2) study drug administered no more than 10 min prior to exercise (5 min target), (3) conducted exercise of moderate to high intensity for at least 30 min and no longer than 75 min, and (4) achieved a target heart rate of 80% of maximum calculated heart rate at least once during session.
  Hypoglycemic event defined as any hypoglycemic event occurring within 30 (+2) min after completion of a qualified exercise session.
Time Frame: Visit 3 (Day 1) and Visit 4 (Day 3 or any day up to Day 29); At each visit, the associated hypoglycemia events were assessed continuously throughout the 30 (+2) minute period following a qualified exercise session.
Population: All randomized subjects in the CRC Phase.
Measure: Number; unit: events/session
Groups:
- CRC Phase: Glucagon RTU With Insulin Pump Reduction: CRC Phase: Glucagon RTU Injection 30 microliters of 0.15 mg injection with 50% reduction in the insulin pump (crossover groups combined)
- CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction: CRC Phase: Vehicle for Glucagon RTU Injection 30 microliters vehicle with 50% reduction in the insulin pump (crossover groups combined)
- CRC Phase: Overall: CRC Phase: Glucagon RTU and/or Vehicle Injection 30 microliters with a 50% reduction in the insulin pump (crossover groups combined)
Arm/Group | CRC Phase: Glucagon RTU With Insulin Pump Reduction | CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | CRC Phase: Overall
Number analyzed (Participants) | 46 | 47 | 48
events/session | 0.02 | 0.19 | 0.11

11. Other Pre Specified Outcome: CRC Phase: Mean Number of Hypoglycemic Events Exercise.
Description: CRC Phase: Mean number of hypoglycemic events associated with the qualified exercise sessions at each CRC Phase visit. With crossover, each subject had 2 exercise sessions; 1 visit and exercise session with each treatment (the combined data are presented in the Overall category) assessed at group level.
  A qualified exercise session is: (1) confirmed blood glucose of 100-180 mg/dL prior to start of exercise, (2) study drug administered no more than 10 min prior to exercise (5 min target), (3) conducted exercise of moderate to high intensity for at least 30 min and no longer than 75 min, and (4) achieved a target heart rate of 80% of maximum calculated heart rate at least once during session.
  A hypoglycemic event defined as any hypoglycemic event occurring within 30 (+2) min after completion of a qualified exercise session.
Time Frame: as for outcome 10
Population: All randomized subjects in the CRC Phase.
Measure: Number; unit: number of events/participant
Arm/Group | CRC Phase: Glucagon RTU With Insulin Pump Reduction | CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | CRC Phase: Overall
Number analyzed (Participants) | 46 | 47 | 48
number of events/participant | 0.02 | 0.19 | 0.21

12. Other Pre Specified Outcome: CRC Phase: Mean Number of Qualified High Intensity Aerobic Exercise Sessions
Description: Mean number of high intensity aerobic exercise sessions at each CRC Phase visit. With crossover, each subject was to have 2 exercise sessions; 1 visit and exercise session with each treatment (the combined data are presented in the Overall category) and assessed at the group level.
  A qualified exercise session was defined as one where (1) confirmed blood glucose of 100-180 mg/dL prior to start of exercise, (2) study drug administered no more than 10 min prior to exercise (5 min target), (3) conducted exercise of moderate to high intensity for at least 30 min and no longer than 75 min, and (4) achieved a target heart rate of 80% of maximum calculated heart rate at least once during session.
Time Frame: Visit 3 (Day 1) and Visit 4 (Day 3 or any day up to Day 29); At each visit, the number of qualified exercise sessions that occurred.
Population: All randomized subjects in the CRC Phase.
Measure: Number; unit: mean number of sessions/participant
Arm/Group | CRC Phase: Glucagon RTU With Insulin Pump Reduction | CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | CRC Phase: Overall
Number analyzed (Participants) | 46 | 47 | 48
mean number of sessions/participant | 1 | 1 | 1.94

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent Form through the followup visit (week 12)
Description: Adverse events were reported and summarized separately for the 2 phases of the study (CRC Phase and Outpatient Phase).
Groups:
- CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction: CRC Phase: 2-arm randomized double-blind crossover, Vehicle for Glucagon RTU Injection 30 microliters vehicle with 50% reduction in insulin pump
- Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction: Outpatient Phase: 3-arm randomized comparison (2-arm double-blind, 1-arm open-label), Vehicle for Glucagon RTU Injection 30 microliters vehicle with 50% reduction in insulin pump (double-blind arm)
Arm/Group | CRC Phase: Glucagon RTU With Insulin Pump Reduction | CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47 | 0/16 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47 | 0/16 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 27/46 | 30/47 | 14/16 | 12/14 | 12/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CRC Phase: Glucagon RTU With Insulin Pump Reduction (N=46) | CRC Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction (N=47) | Outpatient Phase: Glucagon RTU With Insulin Pump Reduction (N=16) | Outpatient Phase: Vehicle for Glucagon RTU With Insulin Pump Reduction (N=14) | Outpatient Phase: Glucagon RTU Without Insulin Pump Reduction (N=14)
Injection site pain (General disorders) | 15 | 18 | 6 | 8 | 3
Injection site discomfort (General disorders) | 4 | 1 | 1 | 1 | 1
Injection site irritation (General disorders) | 1 | 3 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 3 | 0 | 1 | 0
Injection site paresthesia (General disorders) | 0 | 1 | 1 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Application site rash (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 2
Abdominal distension (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Decreased appetiate (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Anhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03841526/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT03841526/SAP_001.pdf